CLINICAL TRIAL: NCT04421716
Title: Phase I Clinical Trial Testing the Bioavailability of Phytonutrients, Curcumin and Ursolic Acid
Brief Title: Testing the Bioavailability of Phytonutrients, Curcumin and Ursolic Acid
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20190940H
Record Dates: First submitted 2020-05-21; First posted 2020-06-09 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Bioavailability of Phytonutrients
MeSH Terms: interventions — Ursolic Acid; Curcumin

STUDY DESIGN:
Intervention Model Description: Cohort 1 and 2 will receive either UA or CURC and Cohort 3 will receive a combination of UA and CURC. Subjects initially enrolled in Cohorts 1 and 2 may have the option to continue in Cohort 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ursolic Acid (Experimental): Administration of Ursolic Acid twice a day for 2 weeks
  Interventions: Drug: Ursolic Acid
- Curcumin (Experimental): Administration of Curcumin twice a day for 2 weeks
  Interventions: Drug: Curcumin
- Ursolic Acid and Curcumin (Experimental): Administration of Ursolic Acid and Curcumin. If subjects from Cohort 1 or 2 wish to continue in the study, they will undergo a washout period of at least 4 weeks before participating in Cohort 3
  Interventions: Drug: Ursolic Acid; Drug: Curcumin

INTERVENTIONS:
Drug: Ursolic Acid — Ursolic Acid 150mg
  Arms: Ursolic Acid; Ursolic Acid and Curcumin
Drug: Curcumin — Curcumin 600mg
  Arms: Curcumin; Ursolic Acid and Curcumin

SUMMARY:
The primary objective of this research is to investigate the bioavailability of curcumin (CURC) and ursolic acid (UA) in a phase I clinical trial in healthy men and obtain biological material for bioavailability analysis.

DETAILED DESCRIPTION:
Once a subject is consented and assigned to a cohort, the subject may undergo a digital rectal exam (DRE) and rectal swab fecal collection and provide research blood (including CBC and CMP safety labs) and urine. Medical history data will be collected and reviewed. The PI and/or study staff will provide supplement administration and supplement diary education prior to the subject starting their dose of UA, CURC, or UA and CURC combination. Pharmacokinetic (PK) and pharmacodynamic (PD) assessments will be collected at pre-dose and 6 and 24 hours after the first dose. Urine will also be collected at pre dose and 24 hours post dose. The dosing period will be for a total of 2 weeks (± 3 days). On the last day of dosing, subjects will attend a research only visit at which the subject may undergo a digital rectal exam (DRE) and rectal swab fecal collection and provide research blood and urine. At this time, the subject's supplement diary will be reviewed and a safety/AE assessment will be completed. In addition, research CBC and CMP safety labs will be collected. If a subject initially enrolled in Cohort 1 or 2 decides to continue in Cohort 3, the subject will undergo a wash out period of at least 4 weeks and repeat all study procedures for Cohort 3.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give informed consent
* Be men age 18 or older
* Able to stop supplements

Exclusion Criteria:

* Unable to give informed consent
* Age < 18
* Woman
* Prisoners
* Diagnosed cancer
* Unable to swallow pills
* Unable to stop supplements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Number, frequency, duration, and relation of toxicity events | Baseline to 2 weeks
  Safety will be compared to evaluate the number, frequency, duration, and relation of toxicity events to CURC and UA, as defined by the Common Terminology Criteria for Adverse Events (CTCAE) v 4.03.
Peak serum concentration | Baseline to 2 weeks
  Dose response curve representing the pharmacokinetic parameter peak serum concentration (Cmax) of ursolic acid, curcumin, and their metabolites will be graphed.
Time to reach peak serum concentration | Baseline to 2 weeks
  The pharmacokinetic parameter, the area under the curve (Tmax) representing the time it takes to reach Cmax of ursolic acid, curcumin, and their metabolites will be graphed.
Half-life | Baseline to 2 weeks
  The pharmacokinetic parameter, half-life of ursolic acid, curcumin, and their metabolites will be graphed.

SECONDARY OUTCOMES:
Microbiome Alpha Diversity | Baseline to 2 weeks
  Number of bacteria collected from rectal culture sample will be assessed before and after each exposure
Microbiome Beta Diversity | Baseline to 2 weeks
  Proportions of bacteria collected from rectal culture sample will be assessed before and after each exposure
Metabolite Panels | Baseline to 2 weeks
  Metabolite panels will be placed into quartiles and compared to predicted function from the bioinformatics tool Phylogenetic Investigation of Communities by Reconstruction of Unobserved States (PICRUSt) software.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Liss, MD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified data will be available upon request following study completion for approx. 1 year.
Access Criteria: Access available upon request.